CLINICAL TRIAL: NCT06667765
Title: A Randomized, Placebo-Controlled, Double-Blinded Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of RPT1G After Single and Multiple Doses in Healthy Adult Participants
Brief Title: A Study of RPT1G After Single and Multiple Doses in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Remedy Plan, Inc. (Industry)
Collaborators: Remedy Plan Australia Pty. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RPT1G
Record Dates: First submitted 2024-10-30; First posted 2024-10-31 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-05

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- RPT1G Single ascending dose (SAD) cohort (Experimental): All participants will receive single oral dose of RPT1G or placebo in fasted state
  Interventions: Drug: RPT1G; Drug: Placebo
- RPT1G Multiple ascending dose (MAD) cohort (Experimental): All participants will receive twice daily oral doses of RPT1G or placebo in a fasted state for 5 days
  Interventions: Drug: RPT1G; Drug: Placebo

INTERVENTIONS:
Drug: RPT1G — Dose formulation- Oral capsule
Drug: Placebo — Dose formulation- Oral capsule

SUMMARY:
This is a first-in-human (FIH), randomized, double-blind, placebo-controlled, single and multiple dose study with staggered dose escalations in healthy participants.

DETAILED DESCRIPTION:
Single-Ascending Dose (SAD) Cohorts: Cohorts 1-4:

Up to 32 participants will be enrolled in this arm. On Day 1, all participants will receive a single oral dose of RPT1G or placebo, in the fasted state, as well as post-dose safety, PK, and PD assessments up to Day 4 (72 hours post-dose).

Multiple-Ascending Dose (MAD) Cohorts: Cohorts 5-7:

Up to 18 participants will be enrolled in this arm. On Day 1, all participants will begin twice daily (BID [i.e., every 12 hours]) multiple oral dose administration of RPT1G or placebo in the fasted state for 5 days as well as safety, PK, and/or PD assessments throughout the study intervention administration period and up to Day 8 (72 hours after last dose).

ELIGIBILITY:
Inclusion Criteria:

1. Must be able to understand and provide written informed consent prior to initiation of study procedures, able to abide by the study restrictions, and remain confined in the research unit as required.
2. Must be ≥ 18 and ≤ 55 years of age, at Screening.
3. Have a body weight ≥ 48 kg (105.6 lbs) and body mass index (BMI) ≥ 18.0 and < 32.0 kg/meter square at Screening, with no clinically significant change in body weight at Check-in as determined by the Investigator.
4. Must be in good health and without clinically significant abnormalities as assessed by review of medical and surgical history, physical examination, vital signs measurement, ophthalmoscopic assessment, and 12-lead ECG at Screening and Check-in as assessed by the Investigator.
5. Laboratory evaluations or laboratory parameters are within the reference range (laboratory parameters outside the reference range may be included only if the Investigator considers that the findings are not clinically significant and agreement by the Sponsor's Medical Monitor is obtained, and inclusion of the participant will not introduce additional risk factors and will not interfere with the study procedures) at Screening and Check-in. One additional repeat laboratory evaluation may be permitted at the Investigator's discretion.
6. Female participants are eligible to enroll and participate in the study if they meet the definition of non-childbearing potential. Women of childbearing potential (WOCBP) can enroll if they have a negative serum pregnancy test result at Screening and agree to comply with the contraception requirements of the protocol. A pregnancy test must also be performed within 72 hours before Day 1 of study dosing.
7. Male participants are eligible to enroll if they agree to comply with the contraception requirements of the protocol.
8. Male participants must agree to not donate sperm during participation in the study starting at Screening and for 3 months following the administration of the last study dose. Female participants must refrain from donating ova and/or breastfeeding during participation in the study and for 30 days following the administration of the last study dose.

Exclusion Criteria:

1. Participant is an employee of the Sponsor, including employees contracted by the Sponsor (i.e., consultants) or an employee of the contract research organization (CRO), or an employee of the site/institution.
2. Any sign or symptom that may indicate an active infection.
3. History of chronic or recurrent infections, or a serious or life-threatening infection within the 6 months prior to Check-in.
4. Hospitalization within 2 months prior to Check-in or major surgical procedure (per Investigator's discretion) of any type within 3 months prior to Check- in.
5. Significant history or clinical manifestation of any metabolic, allergic, autoimmune, dermatological, hepatic, renal, hematological, pulmonary, cardiovascular, gastrointestinal, neurological, ocular, oncologic ( concurrent malignancy or a history of malignancy during the past 5 years, except for basal cell or squamous cell carcinoma-in-situ of the skin that have been successfully excised, or ablated, with no evidence of metastatic disease for 3 years), respiratory, endocrine, or psychiatric disorder, as determined by the Investigator (or designee) that would jeopardize the safety of the individual or the validity of the study results, including any condition that would affect drug absorption, distribution, metabolism, or excretion of drugs (e.g., stomach or intestinal surgery, or gallbladder removal/cholecystectomy; uncomplicated appendectomy and hernia repair will be allowed).
6. Prior treatment with a nicotinamide phosphoribosyltransferase (NAMPT) inhibitor.
7. Use of immunosuppressant therapies or chemotherapy agents or steroids (topical or intranasal steroids for the treatment of hay fever are permissible) within 3 months prior to Screening.
8. History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, unless approved by the Investigator (or designee).
9. Individuals with congenital nonhemolytic hyperbilirubinemia (e.g., suspicion of Gilbert's syndrome based on total and direct bilirubin).
10. Screening or Check-in 12-lead ECG shows:

    1. Prolonged corrected QT interval by Fridericia's method (QTcF) (i.e., QTcF > 450 ms for males and > 470 ms for females)
    2. Other clinically significant abnormalities.
11. Estimated creatinine clearance < 90 mL/min using the Cockcroft-Gault equation at Screening or Check-in.
12. Positive pregnancy test or is lactating (WOCBP) at Screening or Check-in.
13. Has a positive test for human immunodeficiency virus (HIV)-1 or HIV-2 antibodies, hepatitis panel (Hepatitis B surface antibody [HBsAb], Hepatitis B core antibody [HBcAb], and Hepatitis C virus antibody [HCVAb]) or tuberculosis (TB) blood test (e.g., QuantiFERON TB Gold Plus test) at Screening.
14. Use or history of the following: History of alcoholism or drug/chemical abuse within 2 years prior to Check-in. Any use of alcohol within 48 hours of admission to the CRU or positive urine alcohol test result at Check-in. Use of more than 10 tobacco or nicotine containing products (including e-vapor products) per week, or use of any marijuana containing products within 4 weeks prior to Check-in, or positive cotinine at Screening or Check-in. Positive urine drug screen at Screening or Check-in. For each test, one repeat test may be permitted at the Investigator's discretion.
15. Has participated in any investigational study intervention trial in which receipt of an investigational study intervention occurred within 30 days prior to Check-in or 5 half-lives of the investigational intervention's PK, PD, or biological activity (if known), whichever is longer, or is currently participating in another clinical study.
16. Use or intent to use any medications within 30 days or 5 half-lives (whichever is longer) prior to Check-in, unless deemed acceptable by the Investigator (or designee) with agreement by the Medical Monitor.
17. Use or intent to use natural products or nutritional/dietary supplements (including St. John's wort), vitamins, minerals, and phytotherapeutic/herbal/plant-derived preparations within or received within 14 days or 5 half-lives (whichever is longer) prior to Check-in, unless deemed acceptable by the Investigator (or designee) with agreement by the Sponsor's Medical Monitor.
18. Ingestion of Seville/blood oranges, grapefruit, grapefruit hybrids, or marmalade or fruit juice products made from Seville/blood oranges, grapefruit or grapefruit hybrids within 7 days prior to Check-in per the Investigator's discretion.
19. Poor peripheral venous access, receipt of blood products within 2 months prior to Checkin, loss or donation of more than 400mL of blood or blood products during the 8 weeks prior to Check-in, or donation of any blood or blood products during the 2 weeks prior to Check-in.
20. Known history of allergy to any component of study intervention, including excipient(s).
21. Individuals with LFTs > 1.5x ULN.
22. Individuals who, in the opinion of the Investigator (or designee), should not participate in this study.
23. Individuals who have already been enrolled and dosed on this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2024-11-18 (Actual); Primary Completion 2025-05-14 (Actual); Study Completion 2025-05-14 (Actual)

PRIMARY OUTCOMES:
To assess the safety of RPT1G by number of adverse events in accordance with CTCAE V5 | SAD-Day 1 to Day 8 post first dose administration; MAD- Day1 to Day 12 post first dose administration

SECONDARY OUTCOMES:
To evaluate the pharmacokinetics (PK) of RPT1G | Up to 8 days post first dose administration
  Maximum Plasma Concentration (Cmax)
To evaluate the pharmacokinetics (PK) of RPT1G | Up to 8 days post first dose administration
  Time taken for maximum plasma concentration (Tmax)
To evaluate the pharmacokinetics (PK) of RPT1G | Up to 8 days post first dose administration
  Area under the concentration-time curve (AUC)
To evaluate the pharmacokinetics (PK) of RPT1G | Up to 8 days post first dose administration
  Apparent total body clearance (CL/F)
To evaluate the pharmacokinetics (PK) of RPT1G | Up to 8 days post first dose administration
  Terminal half-life (T1/2)
To evaluate the pharmacokinetics (PK) of RPT1G | Up to 8 days post first dose administration
  Apparent total volume of distribution (VZ/F)

CONTACTS AND LOCATIONS:
Locations (1):
- CMAX Clinical Research Pty Ltd, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No